CLINICAL TRIAL: NCT00371228
Title: Delayed Versus Immediate Cord Clamping and Changes in Neonatal Hemoglobin
Brief Title: Timing of Cord Clamping and Neonatal Hemoglobin
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left university
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2005010
Record Dates: First submitted 2006-08-30; First posted 2006-09-01 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Anemia
Keywords: cord clamping; hematocrit; hemoglobin; timing
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Umbilical cord not cut until pulsation stops, in order to provide additional blood to newborn.
  Interventions: Procedure: Delay of umbilical cord clamping
- 2 (No Intervention): Umbilical cord cut soon after birth without waiting for pulsing to stop.

INTERVENTIONS:
Procedure: Delay of umbilical cord clamping — Umbilical cord delayed until pulsation stops.
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether the timing of the clamping of the umbilical cord after delivery has an impact on neonatal hemoglobin and hematocrit, tests that determine the number of red cells in the blood and their ability to carry oxygen. The study hypothesis is that delaying cord clamping until cord pulsation has ceased will increase the neonatal blood volume and thereby increase the hemoglobin and hematocrit.

We propose to recruit 150 women who present for vaginal delivery at Tulsa Regional Medical Center. Half of the women will be randomly assigned to the immediate clamping group, which will entail clamping of the umbilical cord within six seconds of delivery of the fetal shoulders. The other half of the volunteers will be assigned to the delayed clamping group, which will entail clamping the cord after a palpable pulse has ceased, or after 10 minutes. The infants of mothers in both groups will have blood drawn for a hemoglobin and hematocrit at the time of the routine PKU heel stick, usually is performed within 18-24 hours of delivery.

Statistical differences between the blood counts of infants in the control and study groups will be compared using independent samples t tests.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the timing of the clamping of the umbilical cord after delivery has an impact on neonatal hemoglobin and hematocrit, tests that determine the number of red cells in the blood and their ability to carry oxygen. The study hypothesis is that delaying cord clamping until cord pulsation has ceased will increase the neonatal blood volume and thereby increase the hemoglobin and hematocrit.

As the communication between the placenta and fetus, the umbilical cord provides oxygen and nutrients until the time of delivery. Even after delivery, placental respiration continues for a short time and the newborn infant continues to receive blood from the placenta until physiologic closure of the cord vessels terminates the transfusion. While most term infants can tolerate variations in blood volume, those who are compromised by prematurity, cesarean delivery or cord compression in utero may require blood transfusions if the cord is clamped before pulmonary perfusion is established. Delayed cord clamping is believed to provide a greater supply of blood to perfuse the lungs without robbing blood from the other organs.

In uncomplicated vaginal deliveries the umbilical cord traditionally has been clamped immediately after delivery, more for the doctor's convenience than for any consideration regarding the health of the infant. Both immediate and delayed cord clamping are accepted as routine standard of care at delivery, depending on the circumstances. However, some clinicians and researchers have suggested that by delaying the clamping of the umbilical cord, the placental transfusion to the newborn is maintained, optimizing blood volume and hemostasis.

Several European research studies have suggested that delayed cord clamping increases newborn hemoglobin and hematocrit. However, these studies were not performed under properly controlled conditions and thus have failed to gain general acceptance.

We propose to recruit 150 women who present for vaginal delivery at Tulsa Regional Medical Center. We believe this number of volunteers is possible to enroll in the allotted five months for data collection. A power analysis for this sample size was performed by Dr. Mark Payton, professor of statistics at the OSU Stillwater campus. He estimated that a difference of 0.3 standard deviations has a power of just over 95%.

OSU medical students will explain the study and recruit patient volunteers during routine third trimester prenatal care visits at the OSU OB/Gyn resident clinic at Houston Parke. Study investigators Drs. Beal and Carnett will determine the eligibility of those patients who agree to participate. The ethnic mix of the resident clinic population is not available because race information is not routinely entered in the MegaWest Practice Management Program currently in use.

When a volunteer presents for delivery, the resident in charge of the labor and delivery unit will remind the patient of her previous consent to participate and assign her to either the control group or the study group in an alternating fashion. Women who have agreed to participate in the study will have an identifying mark on their prenatal records which are sent from the clinic. In the control group, the umbilical cord will be clamped immediately after delivery. In the study group, the umbilical cord will be clamped once cord pulsation ceases. Patients also will be advised at this time that they can withdraw from the study at any time, regardless of the reason. The physician making group assignments and performing deliveries on a given day may not be one of the study investigators.

The inability to mask the patients and study personnel will not affect the outcome of the study as strict guidelines regarding the timing of cord clamping will be applied. Immediate clamping will entail clamping of the umbilical cord within six seconds of delivery of the fetal shoulders. Delayed clamping will be performed by clamping the cord after a palpable pulse has ceased, or after 10 minutes. Cord pulsation generally stops within two minutes of delivery. The physician performing the delivery will determine when cord pulsation stops and the clamp times, immediate or delayed will be recorded by delivery room personnel who routinely record times of delivery of infant, delivery of placenta, infant weight and APGARs. Therefore, prior knowledge of group assignment will not affect the behavior of the patient or the physician at the time of delivery.

The infants of mothers in both groups will have blood drawn for a hemoglobin and hematocrit at the time of the routine PKU heel stick. There will be no additional heel sticks to collect blood. The PKU test usually is performed within 18-24 hours of delivery. All infant study data will be collected at this time and no further blood draws will be necessary. The total amount of blood drawn from the baby will be approximately 8-10 drops, or about two teaspoons, which will include blood for the PKU test and the study tests. The results of the blood tests will then be analyzed and compared between the two groups. This comparison will also involve analysis of the mothers' admitting hemoglobin and hematocrit, blood type and demographic data, including age and smoking history, to look for possible exclusion or confounding factors. Maternal blood is routinely tested at the time of admission for blood type, hemoglobin and hematocrit. This involves the collection of approximately two test tubes of blood. No additional testing or blood collections will be performed on participating mothers other than those routinely done.

There are no increased risks to mothers or their infants who agree to participate in the study. Likewise, there are no direct benefits to participation to either mothers or babies aside from the contribution their participation makes in furthering medical knowledge. Adverse events and serious adverse events will be recorded and reported to the IRB under the policies and procedures provided by OSUCHS.

Our tentative timetable is to recruit 25 patients per month so that the data collection can be completed within five months. Tulsa Regional typically delivers about 1,000 babies monthly. Approximately 23 percent of these deliveries are cesarean sections. Of the remaining deliveries, it is reasonable to estimate that 25 patients per month could be recruited to the study.

The study population will include 150 women and their newborn infants delivered at Tulsa Regional Medical Center. Mothers must be between the ages of 18 and 34 and be full term, 37 to 41 weeks, with a singleton pregnancy at the time of delivery. Women will be excluded from the study if their delivery is complicated by non-reassuring fetal heart tones, preeclampsia, eclampsia, chronic hypertension, meconium-stained amniotic fluid, fetal anomalies or any other condition which could require immediate newborn evaluation by nursery personnel at the time of delivery. Infants requiring operative delivery by forceps or vacuum also will be excluded.

Analysis Statistical differences between the blood counts of infants in the control and study groups will be compared using independent samples t tests.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women and their newborn infants delivered at Tulsa Regional Medical Center,
* between the ages of 18 and 34,
* full term (37 to 41 weeks),
* singleton pregnancy at the time of delivery

Exclusion Criteria:

* Delivery complicated by non-reassuring fetal heart tones,
* preeclampsia,
* eclampsia,
* chronic hypertension,
* meconium-stained amniotic fluid,
* fetal anomalies or
* any other condition which could require immediate newborn evaluation by nursery personnel at the time of delivery. Infants requiring operative delivery by forceps or vacuum also will be excluded.

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2006-09 (Estimated); Primary Completion 2009-06 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
hemoglobin | day of birth

CONTACTS AND LOCATIONS:
Overall Officials: John M. Beal, D.O., Principal Investigator — Oklahoma State University Center for Health Sciences
Locations (1):
- OSU Houston Center, Tulsa, Oklahoma, United States